CLINICAL TRIAL: NCT03500341
Title: Oxygen Reserve Index (ORi) Validation of INVSENSOR00014
Status: Terminated | Type: Interventional
Why Stopped: The data from the study showed good trending of Delta ORi and Delta PaO2. The study was stopped before full enrollment as a newer version of ORi was developed.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19193
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00014 sensor
  Interventions: Device: INVSENSOR00014

INTERVENTIONS:
Device: INVSENSOR00014 — Noninvasive pulse oximeter sensor

SUMMARY:
The Oxygen Reserve Index (ORi) is a reference that could help clinicians with their assessments of normoxic and hyperoxic states by scaling the measured absorption information between 0.00 and 1.00. An ORi of 0.00 corresponds to PaO2 values of 100mmHg and below and an ORi of 1.00 corresponds to PaO2 values of 200mmHg and above.) In this study, the PaO2 is varied by controlling the concentration of oxygen the study volunteer breathes. The ORI device measurement is analyzed by comparing it to the PaO2 measurements from blood samples from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate greater than or equal to 45 bpm and less than or equal to 85 bpm.
* Carbon monoxide (CO) value less than or equal to 2.0% fractional carboxyhaemoglobin (FCOHb)
* Subject has a physical status of American Society of Anesthesiology Class 1 (ASA I, Healthy subjects without any systemic disease at all.) American Society of Anesthesiology Class 2 (ASA II, subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure less than or equal to 140 mmHg and Diastolic Blood Pressure less than or equal to 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (smoking includes e-cigarette use)
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has open wounds, inflamed tattoos or piercings or any visible healing wounds.
* Subject experiences frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse or uses recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last year.
* Subject has any chronic bleeding disorders (i.e. hemophilia)
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer).
* Subject has a chronic neurological disease (i.e. multiple sclerosis, Huntington's disease).
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subjects' level of consciousness.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator).
* Subject has Wolff-Parkinson-White Syndrome or Stokes - Adams syndrome.
* Subject who has taken anticoagulant medications within the last 30 days.
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ear nose or throat (ENT) surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has donated blood within the last 2 weeks.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has had a concussion within the past 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent Diabetes or uncontrolled hypertension.
* Subject has given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization, or had a cesarean section (C-section) within the past 6 months.
* Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours of the study.
* Discretion of investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 enrolled participants, 16 met inclusion criteria and proceeded to the study. The remainder of the enrolled participants include screen failures and subjects that did not proceed due to time constraints.
Period: Overall Study
Arm/Group | Test Subject
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawn prior to Completion | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Subject
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 0
  18 to 50 years old | 14
  > 50 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4
  Black or African American | 3
  Native American | 2
  Hispanic | 3
  Asian or Pacific Islander | 2

OUTCOME MEASURES:

1. Primary Outcome: Specificity, Sensitivity, and Concordance for the ORi Measurement System as Compared to PaO2
Description: This study reports ORi specificity, sensitivity and concordance for Masimo's ORi measurement system as compared to PaO2 from blood samples.
Time Frame: 1-5 hours per subject
Population: Sufficient number of cases to meet sample size criteria for assessing outcomes was not achieved. The protocol required a minimum of 22 completed subjects. This study was not able to meet this target and therefore the specificity, sensitivity and concordance for Masimo's ORi measurement system could not be defined (primary outcome measure).
Arm/Group | Test Subject
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | Test Subject
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03500341/Prot_SAP_000.pdf